CLINICAL TRIAL: NCT06582719
Title: Evaluating the Efficacy of GPT-based Nutrition and Diabetic Counseling in Gestational Diabetes Management: A Randomized Controlled Trial (AIM-GDM)
Acronym: AIM-GDM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-16035
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutritional Counseling plus AI Intervention (Experimental)
  Interventions: Device: GPT-based counseling; Other: Nutritional Counseling
- Nutritional Counseling (Active Comparator)
  Interventions: Other: Nutritional Counseling

INTERVENTIONS:
Device: GPT-based counseling — AI-based counseling provided to the patient, accessible on their smartphone device at the time of Gestational Diabetes diagnosis
  Arms: Nutritional Counseling plus AI Intervention
Other: Nutritional Counseling — Standard Nutritional Counselling provided by a registered dietician at the time of Gestational Diabetes diagnosis

SUMMARY:
The purpose of this study is to assess whether an AI based counseling service can be beneficial for patients to assist in management of gestational diabetes.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) affects approximately 6-9% of pregnancies globally, posing significant risks to both maternal and neonatal health. Standard management includes dietary counseling, glucose monitoring, and insulin therapy when necessary. However, the rising prevalence of GDM and limited healthcare resources necessitate innovative solutions to supplement traditional care. Generative Pre-trained Transformers (GPTs), a type of large language model (LLM), offer personalized, real-time counseling and support. Recent advancements in AI have shown promise in various healthcare applications, but the efficacy of GPT-based counseling in GDM management remains underexplored. This study builds on preliminary evidence suggesting that AI can enhance patient engagement and outcomes, aiming to validate these findings in a controlled trial.

The integration of AI, specifically GPTs, into healthcare can revolutionize patient management by providing continuous, tailored support. This study aims to evaluate whether GPT-based counseling can improve glycemic control and patient satisfaction in GDM management, compared to traditional counseling alone. By placing AI within the context of prenatal care, this research seeks to address gaps in current GDM management practices and offer scalable, personalized solutions.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45
* Diagnosed with GDM in pregnancy
* Able to use a smartphone
* Fluent in English or Spanish

Exclusion Criteria:

* Pre-existing diabetes
* High-risk pregnancies due to other medical conditions
* Inability to consent
* Non-English and/or Non-Spanish speakers
* No smartphone access

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnant women are elligible
Enrollment: 80 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Birth weight at time of Delivery | Within 12 hours of delivery
  Newborns will be weighed within 12 hours of the time of delivery. Birth weights will be summarized and reported by study group using basic descriptive statistics. Higher birth weights have been associated with Gestational Diabetes Mellitus (GDM) and increased risk of perinatal complications.

SECONDARY OUTCOMES:
Rate of Neonatal Intensive Care Unit (NICU) admissions | Within 12 hours of delivery
  Rate of NICU admission will be expressed as the percentage of newborns who were admitted to the NICU within 12 hours of delivery. Rates will be summarized and reported by study group using basic descriptive statistics. Increased admissions to the NICU are associated with less favorable perinatal outcomes.
Rate of Cesarean Section | Within 12 hours of delivery
  Rate of Cesarean Section will be expressed as the percentage of patients who delivered via Cesarean section. Rates will be summarized and reported by study group using basic descriptive statistics. Patients with GDM are more likely to need Cesarean sections leading to less favorable perinatal outcomes for the newborn.
Rate of Progression to medication requirements | At the time of delivery
  The rate of progression to medication requirements for GDM will be assessed as the percentage of patients who are administered either insulin or oral hypoglycemic at the time of delivery. Rates will be summarized and reported by study group using basic descriptive statistics. Higher rates of progression to medications are associated with increased hyperglycemia and less favorable perinatal outcomes in general.
Rate of Shoulder Dystocia | Within 12 hours of delivery
  Rate of Shoulder Dystocia will be expressed as the percentage of patients who have been diagnosed with should dystocia within 12 hours of delivery. Rates will be summarized and reported by study group using basic descriptive statistics. GDM is a risk factor for shoulder dystocia and higher rates of shoulder dystocia are associated with increased perinatal complications.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Mastrogiannis, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander GR, Himes JH, Kaufman RB, Mor J, Kogan M. A United States national reference for fetal growth. Obstet Gynecol. 1996 Feb;87(2):163-8. doi: 10.1016/0029-7844(95)00386-X. PMID 8559516
- [Background] Centers for Disease Control and Prevention (CDC). (2022). National Diabetes Statistics Report